CLINICAL TRIAL: NCT00025636
Title: A Randomized Trial Of BEAM Plus PBSCT Versus Single Agent High-Dose Therapy Followed By BEAM Plus PBSCT In Patients With Relapsed Hodgkin's Disease
Brief Title: Combination Chemotherapy and Peripheral Stem Cell Transplant in Treating Patients With Relapsed Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: German Hodgkin's Lymphoma Study Group (Other)
Collaborators: European Organisation for Research and Treatment of Cancer - EORTC (Network); EBMT Solid Tumors Working Party (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068981; GHSG-HD-R2; EBMT-GHSG-HD-R2; EORTC-20011
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2007-06

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease | interventions — Filgrastim; Carmustine; Cisplatin; Cyclophosphamide; Cytarabine; Dexamethasone; Etoposide; Melphalan; Methotrexate; Vincristine; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: carmustine
Drug: cisplatin
Drug: cyclophosphamide
Drug: cytarabine
Drug: dexamethasone
Drug: etoposide
Drug: melphalan
Drug: methotrexate
Drug: vincristine sulfate
Procedure: bone marrow ablation with stem cell support
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Peripheral stem cell transplant may allow the doctors to give higher doses of chemotherapy drugs and kill more cancer cells. It is not yet known which combination chemotherapy regimen given before peripheral stem cell transplant is more effective in treating relapsed Hodgkin's lymphoma.

PURPOSE: This randomized phase III trial is comparing different regimens of combination chemotherapy followed by peripheral stem cell transplant to see how well they work in treating patients with relapsed Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of induction chemotherapy followed by combination chemotherapy and autologous peripheral blood stem cell transplantation with or without high-dose sequential chemotherapy in terms of freedom from treatment failure in patients with relapsed Hodgkin's lymphoma.
* Compare the toxicity of these regimens in these patients.
* Compare the complete remission/unconfirmed complete remission rate at 3 months, relapse-free survival, and overall survival of patients treated with these regimens.
* Compare the frequency of severe toxic effects and secondary neoplasia in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center, type of relapse (early first relapse [remission duration 3-12 months] vs late first relapse [remission duration more than 12 months] vs second relapse without prior high-dose chemotherapy salvage [remission duration after salvage at least 3 months]), disease status at relapse (stage I or II vs stage III or IV), age (18 to 49 vs 50 to 60), and response after 2 courses of study induction chemotherapy (complete remission vs partial remission vs no change).

All patients receive induction chemotherapy comprising dexamethasone IV over 30 minutes on days 1-4 and 15-18, cisplatin IV continuously over 24 hours on days 1 and 15, cytarabine IV over 3 hours every 12 hours on days 2 and 16, and filgrastim (G-CSF) subcutaneously (SC) once daily on days 5-12 and days 19-26. Patients with complete remission (CR), unconfirmed CR, partial remission, or no change are randomized to one of two treatment arms.

* Arm I: Patients receive BEAM chemotherapy comprising carmustine IV over 30 minutes and melphalan IV over 30 minutes on day 37 and etoposide IV over 30 minutes every 12 hours and cytarabine IV over 30 minutes every 12 hours on days 37-40. Patients also receive G-CSF SC twice daily beginning on day 41 and continuing until blood counts recover. Autologous peripheral blood stem cells (PBSCs) are reinfused on day 42.
* Arm II: Patients receive high-dose cyclophosphamide IV over 8 hours on day 37, high-dose methotrexate IV over 6 hours and high-dose vincristine IV on day 51, and high-dose etoposide IV over 8 hours on days 58-61. Patients then receive BEAM chemotherapy comprising carmustine IV over 30 minutes and melphalan IV over 30 minutes on day 80 and etoposide IV over 30 minutes every 12 hours and cytarabine IV over 30 minutes every 12 hours on days 80-83. Patients also receive G-CSF SC once on days 38 and 62 and twice daily beginning on day 84 and continuing until blood counts recover. Autologous PBSCs are reinfused on day 85.

Patients with residual lymphoma at 100 days after completion of BEAM chemotherapy may receive radiotherapy.

Patients are followed at 100 days after PBSC transplantation, every 3 months for 2 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A minimum of 220 patients (110 per treatment arm) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Hodgkin's lymphoma
* Early or late first relapse

  * Complete or partial remission for at least 3 months after completion of prior COPP/ABVD, COPP/ABV/IMEP, MOPP/ABV, ABVD, BEACOPP, or other polychemotherapy regimen with or without radiotherapy
  * No prior salvage therapy OR
* Second relapse

  * Any prior salvage therapy
  * No prior high-dose chemotherapy

PATIENT CHARACTERISTICS:

Age:

* 18 to 60

Performance status:

* Karnofsky 70-100% OR
* ECOG 0-2

Life expectancy:

* More than 3 months with treatment

Hematopoietic:

* Absolute neutrophil count at least 2,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Not specified

Renal:

* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No uncontrolled hypertension (diastolic blood pressure greater than 115 mm Hg)
* No unstable angina
* No New York Heart Association class III or IV heart disease (congestive heart failure)
* No myocardial infarction within the past 6 months
* No uncontrolled atrial or ventricular cardiac arrhythmias

Pulmonary:

* No chronic pulmonary disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No active infection
* No poorly controlled diabetes
* No cerebral disorder
* No other concurrent malignancy except adequately treated basal cell skin cancer or cervical intraepithelial neoplasia
* No significant non-malignant disease
* No psychiatric, addictive, or other disorder that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* No other concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* Not specified

Other:

* At least 6 months since prior coronary angioplasty
* No other concurrent investigational drugs
* No concurrent non-steroidal anti-inflammatory drugs, salicylate, sulfonamide, trimethoprim, allopurinol, aminoglycoside, amoxicillin, or probenecid during high-dose methotrexate administration

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2001-07

PRIMARY OUTCOMES:
Efficacy at 3 months
Toxicity at 3 months

SECONDARY OUTCOMES:
Complete remission at 3 months
Relapse-free survival at 3 months
Overall survival at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Engert, MD — Medizinische Universitaetsklinik I at the University of Cologne; J. W. Baars, MD, PhD — The Netherlands Cancer Institute; Norbert Schmitz, MD, PhD — Asklepios Klinik St. Georg
Locations (44):
- Belgium (4):
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - Algemeen Ziekenhuis Sint Lucas, Ghent
- University Hospital Rebro, Zagreb, Croatia
- Rigshospitalet - Copenhagen University Hospital, Copenhagen, Denmark
- Germany (27):
  - Charite - Campus Charite Mitte, Berlin
  - Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Charite - Campus Virchow Klinikum, Berlin
  - Medizinische Poliklinik, Bonn
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - Staedtisches Klinikum Dessau, Dessau
  - Universitaetsklinikum Essen, Essen
  - Evangelisches Krankenhaus Essen Werden, Essen
  - Klinik Fuer Innere Medizin, Hematology/Oncology, Ernst Moritz Armdt Universitaet, Greifswald
  - Martin Luther Universitaet, Halle
  - Asklepios Klinik St. Georg, Hamburg
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Evangelische Krankenhaus Hamm, Hamm
  - Krankenhaus Siloah - Medizinische Klinik II, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Medizinische Universitaetsklinik und Poliklinik, Heidelberg
  - St. Bernward Krankenhaus, Hildeshem
  - Universitaetsklinikum des Saarlandes, Homburg
  - Clinic for Bone Marrow Transplantation and Hematology and Oncology, Idar-Oberstein
  - Klinikum der Friedrich-Schiller Universitaet Jena, Jena
  - Staedtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck
  - Krankenhaus Muenchen Schwabing, Munich
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Diakonie Klinikum Stuttgart, Stuttgart
  - Dr. Horst-Schmidt-Kliniken, Wiesbaden
- Netherlands (8):
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academisch Medisch Centrum at University of Amsterdam, Amsterdam
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
  - Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen
  - Maxima Medisch Centrum - Veldhoven, Veldhoven
- Maria Sklodowska-Curie Memorial Cancer Center and Institute of Oncology, Warsaw, Poland
- Hospitais da Universidade de Coimbra (HUC), Coimbra, Portugal
- UniversitaetsSpital Zuerich, Zurich, Switzerland

REFERENCES:
- [Derived] Brockelmann PJ, Muller H, Casasnovas O, Hutchings M, von Tresckow B, Jurgens M, McCall SJ, Morschhauser F, Fuchs M, Borchmann P, Moskowitz CH, Engert A. Risk factors and a prognostic score for survival after autologous stem-cell transplantation for relapsed or refractory Hodgkin lymphoma. Ann Oncol. 2017 Jun 1;28(6):1352-1358. doi: 10.1093/annonc/mdx072. PMID 28327958